CLINICAL TRIAL: NCT03447639
Title: A Randomized Trial of Betadine Bladder Irrigations vs. Standard of Care Prior to Indwelling Catheter Removal to Reduce Bacteriuria and Catheter-Associated Urinary Tract Infections
Brief Title: Betadine Bladder Irrigations vs. Standard of Care Prior to Indwelling Catheter Removal
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Patient Enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Jay Hollander MD, Attending Urologist, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-001
Record Dates: First submitted 2018-02-08; First posted 2018-02-27 (Actual); Results first posted 2019-04-24 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Catheter; Infection (Indwelling Catheter); Catheter Infection; Catheter-Related Infections; Catheter Bacteraemia; Urinary Tract Infections
Keywords: Catheter associated UTI; Povidine iodine; Bladder Irrigation
MeSH Terms: conditions — Infections; Catheter-Related Infections; Urinary Tract Infections | interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: 2 arm parallel study with 1 to 1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Povidone-Iodine Irrigation (Experimental): Bladder irrigation with 2% povidine-iodine irrigation immediately prior to catheter removal
  Interventions: Drug: Povidone-iodine irrigation
- Standard of Care (No Intervention): Catheter removal with no bladder irrigation

INTERVENTIONS:
Drug: Povidone-iodine irrigation — Single dose, 60 cc of 2% povidone-iodine indwelling for 10 minutes prior to catheter removal using aseptic technique
  Other Names: Betadine
  Arms: Povidone-Iodine Irrigation

SUMMARY:
Over the last decade, there has been great emphasis on reducing the incidence of hospital-acquired infections, including catheter-associated UTI (CAUTI). This study will evaluate the effectiveness of Betadine irrigation solution (2% povidone-iodine) instilled into the bladder immediately prior to indwelling catheter removal to decrease the risk of subsequent bacteriuria, leading to decreased rates of NHSN defined CAUTI.

DETAILED DESCRIPTION:
Indwelling urinary catheters are routinely used in the care of hospitalized patients for a variety of reasons, including monitoring of urine output in critically ill patients, relief of urinary obstruction, and prevention of contamination of decubitus ulcers. Bacteriuria increases by 3-10% each day a catheter is left in place, meaning that by 30 days, generally 100% of patients with indwelling catheters will have bacteria in their urine. The majority of these people do not have urinary tract infections (UTIs), they are merely colonized and do not require treatment.

To define a standard (and ultimately to compare hospitals against each other), a surveillance definition for CAUTI has been developed by the National Healthcare Safety Network (NHSN). While useful for surveillance, the definition does not correlate with clinical UTIs, leading to over diagnosis and over-reporting of UTIs (in other words, those with merely bladder colonization being diagnosed as having a UTI). Despite continuing progress in standard methods of reducing infection rates (including decreasing the number of catheters inserted, ensuring proper catheter maintenance, and removing catheters when no long necessary) there continue to be unacceptably high rates of CAUTIs.

A single dose of povidone-iodine prior to catheter removal seems a novel and promising practice for several reasons. First, we suspect it will be helpful in reducing rates of NHSN defined CAUTI, as these are still diagnosed for 2 days after the catheter is removed. Second, using multiple doses of povidone-iodine would be inadvisable, since we suspect bacteria over time would become resistant even to this antiseptic. Third, we suspect use of an antiseptic is preferable to an antibacterial for preventing further antimicrobial resistance development. Finally, use of this method, as opposed to the suggested use of systemic antibiotics at time of removal, is potentially preferable from the downstream standpoint of less antimicrobial resistance and reduced risk of Clostridium difficile infection.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and the willingness and ability to comply with all aspects of study requirements
2. Male
3. Inpatients ≥ 18 years of age with an indwelling catheter in place for at least 5 days with a plan for removal

Exclusion Criteria:

1. Patients planned for discharge with an indwelling catheter in place
2. Patients unable to report urinary symptoms accurately
3. Patients with hyper-sensitivity or allergic reaction to Betadine, iodine, shellfish or other related compounds
4. Clinical signs or symptoms of urinary tract infection at the time of consent
5. Patients currently being treated for UTI
6. Patients currently taking any antibiotic medication, other than vancomycin, linezolid, daptomycin, clindamycin, or metronidazole.
7. Patients already taking medications known to potentially irritate the bladder, such as, but not limited to, cyclophosphamide, ifosfamide, and other chemotherapeutic agents
8. Patients with history of bladder cancer, pelvic radiation or interstitial cystitis
9. Patients unable to comply with study requirements
10. Any other condition which, per investigators' judgment, may increase patient risk and/or impede the reliability of study data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hollander, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the inpatient units of the hospital.
Period: Overall Study
Arm/Group | Povidone-Iodine Irrigation | Standard of Care
Started | 0 (No patients were randomized to the Povidone-Iodine irrigation arm) | 3 (3 patients were randomized to the Standard of Care arm.)
Completed | 0 (No patients were randomized to the Povidone-Iodine irrigation arm) | 1 (2 patients were withdrawn because their catheters had to be re-inserted.)
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: No patients were randomized to the Povidone-Iodine arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Povidone-Iodine Irrigation | Standard of Care | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants] — Collected from the medical record
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 3 | 3
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 3 | 3
Presence of urinary tract infection [Count of Participants; unit: Participants] — Positive urinary tract infection (UTI) is defined as a positive urinalysis, culture and patient reported UTI symptoms.
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis of Urinary Tract Infection (UTI)
Description: Per NHSN defined catheter associated UTI (CAUTI) criteria
Time Frame: 48-72 hours after catheter removal
Population: Patients with an indwelling catheter meeting the study eligibility criteria
Arm/Group | Povidone-Iodine Irrigation | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Diagnosis of UTI at 7 Days
Description: Per National Healthcare Safety Network (NHSN) defined CAUTI criteria
Time Frame: 7 days after catheter removal
Population: Study terminated due to low enrollment
Arm/Group | Povidone-Iodine Irrigation | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Diagnosis of UTI at 28 Days
Description: Per NHSN defined CAUTI criteria
Time Frame: 28 days after catheter removal
Population: Study terminated due to low enrollment
Arm/Group | Povidone-Iodine Irrigation | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days; from study enrollment through the study completion
Description: No patients were enrolled in the povidone-iodine arm of the study
Arm/Group | Povidone-Iodine Irrigation | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT03447639/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03447639/ICF_001.pdf